CLINICAL TRIAL: NCT05475418
Title: Pilot Study of Human Adipose Tissue Derived Exosomes Promoting Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Drkailiu
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2022-02

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Adipose tissue derived exosomes — 200-300ml of the subject adipose tissue before centrifugation was collected, and the extracellular vesicles were retained after tissue homogenate and filter screening. The extracellular vesicles were mixed with sterile hydrogel and applied directly to the wound surface, and the wound was covered with an inert protective dressing.

SUMMARY:
This study is a one-arm pilot study. All patients were recruited on an outpatient basis. After screening visits and informed consent was obtained, debridement and photography were performed on the patient's wound surface, and the wound area was measured. Patients in the intervention group were then provided with adipose tissue exosome dressings.200-300ml of the subject adipose tissue before centrifugation was collected, and the extracellular vesicles were retained after tissue homogenate and filter screening. The extracellular vesicles were mixed with sterile hydrogel and applied directly to the wound surface, and the wound was covered with an inert protective dressing.

DETAILED DESCRIPTION:
After giving written informed consent, participants will be followed up once a week during the 2-week lead-in period to confirm that they meet the inclusion criteria.Patients who meet inclusion and exclusion criteria at the end of the induction period will receive treatment twice a week for 4 weeks or until recovery, whichever occurs first.When the observer confirmed that the wound had healed, the patient was followed up for two healing visits within the next 2 weeks.If the evaluator confirms target wound healing at the 4-week confirmatory follow-up, subjects will enter the study follow-up phase, which will be completed at 4 and 6 weeks after the end of the initiation phase.If the target wound did not heal after 6 weeks of treatment, participants completed follow-up at 4 and 6 weeks after the initiation period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 18 to 60, regardless of gender; 2. Full-layer skin wounds on various parts of the body, lasting 4-8 weeks A. For post-amputation wounds, the time between operation and amputation must be more than 30 days; B. If there are wounds >1, select the largest wound as the research target; 3. At the beginning of the induction period, the wound size after debridement was ≥1 and ≤20 cm2; 4. Texas grade 1A, 1B, 1C, 1D, 2A, 2B, 2C or 2D; 5. Ankle-brachial index ≥0.7, including percutaneous oxygen pressure (TcPO2) ≥30 mm hg and skin perfusion pressure ≥30 mm hg; 6. No revascularization procedure or vascular surgery planned within the past or next 30 days; 7. The subject and their family members are willing and able to comply with all prescribed requirements for care and consultation; 8. Subjects have reasonable expectations of completing the study; 9. Subjects completed 2 weeks of initiation and wound reduction was 30%

Exclusion Criteria:

* 1. Signs of gangrene in any part of the torso and limbs of the subject; 2. Written diagnosis of osteomyelitis in any part of the affected limb; 3. Bone tissue at the wound site was exposed; 4. Poor blood glucose control: HbA1c>12% (108 mmol/mol); 5. Subject is receiving kidney dialysis or creatinine >2.5mg/ dL (221mmol/L); 6. The subject has obvious immune deficiency; 7. The subject has suspected tumor or is receiving tumor treatment; 8. Long-term use of steroids or immunosuppressants within the past 3 months or expected use during the study period; 9. During the screening period, subjects have received growth factor therapy, autologous platelet-rich plasma gel, bilayer cell therapy, dermal substitutes, extracellular matrix, etc.

  10. Subject participated in another research device, drug or biological trial within the past 30 days; 11. The wound showed severe symptoms of clinical infection, requiring hospitalization or immediate surgical treatment; 12. The subject has developed deep vein thrombosis within the past 30 days; 13. The subject is pregnant or breastfeeding; 14. The subject has serious mental illness and psychological abnormality; 15. The subject was determined by the attending physician to be unfit for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of wound healing in each group at 4 weeks | 4 weeks
  Percentage of wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Kai Liu, MD,PhD, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu W, Liu T, Zhao Q, Ma J, Jiang J, Shi H. Adipose Tissue-Derived Extracellular Vesicles: A Promising Biomarker and Therapeutic Strategy for Metabolic Disorders. Stem Cells Int. 2023 Dec 26;2023:9517826. doi: 10.1155/2023/9517826. eCollection 2023. PMID 38169960